CLINICAL TRIAL: NCT03829722
Title: Phase II Trial of Radiotherapy, Carboplatin/Paclitaxel and Nivolumab for High Risk HPV-Related Oropharynx Cancer
Brief Title: Radiotherapy, Carboplatin/Paclitaxel and Nivolumab for High Risk HPV-related Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.085; HUM00154941 (Other: University of Michigan)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Oropharynx Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab, Carboplatin/Paclitaxel, Radiotherapy (Experimental): Therapy will continue for 21 weeks total. This includes 4 doses of of nivolumab (240mg/m2) before and concurrent with RT/carboplatin/paclitaxel and 4 adjuvant nivolumab doses (480mg/m2) after the end of RT.
  Interventions: Drug: Nivolumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — Given intravenously (IV), 240 mg every 2 weeks for 4 doses concurrent with radiation therapy (RT). Following completion of RT, 480 mg given every 4 weeks for 4 doses.
  Other Names: Opdivo; BMS-936558; MDX1106; ONO-4538
Drug: Carboplatin — Given IV once per week during radiation therapy (AUC=1).
  Other Names: Paraplatin
Drug: Paclitaxel — Given IV once per week during radiation therapy (30mg/m^2)
  Other Names: Taxol
Radiation: Radiation Therapy — Given 5 days/week for a total of 35 doses (70 gray total).

SUMMARY:
The purpose of this study is to find out if the addition of nivolumab can improve 2 year progression free survival (PFS) as compared to standard of care of fractionated radiation therapy (RT) and carboplatin/paclitaxel in subjects with high risk HPV-related squamous cell carcinoma of the oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate). Fractionated means the radiation will be administered in fragments or parts across multiple days.

DETAILED DESCRIPTION:
PCD details were updated as RECIST is not appropriate for tumor response assessment in this population. Tumor response will be assessed via clinical assessment and PET response (determining progression and location, if any evidence of disease).

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically proven squamous cell carcinoma of the oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate) that is p16 positive by immunohistochemistry or HPV positive by in situ hybridization
* Clinical stage: stage III AJCC 8th edition staging (cT4 or cN3) OR "matted lymph nodes" (defined as 3 LNs abutting one another with loss of intervening fat plane that is replaced with evidence of extracapsular spread)
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination, including documentation of weight within 2 weeks prior to registration;
  * FDG-PET/CT scan for staging and RT plan within 4 weeks prior to registration; Zubrod Performance Status 0-1 within 2 weeks prior to registration;
  * Age ≥ 18;
* CBC/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3; Platelets ≥ 75,000 cells/mm3; Hemoglobin ≥ 9.0 g/dL AST/ALT <3 x ULN
  * Total Bilirubin <1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level < 3 x ULN)
* Serum creatinine within normal institutional limits or a creatinine clearance ≥ 45 mL/min within 2 weeks prior to registration;
* Women of childbearing potential must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study and for five months after the last treatment. A woman of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause. Men receiving nivolumab who are sexually active with WOCBP must agree to use effective contraception throughout their participation in the treatment phase of the study and for seven months after the last treatment.
* Due to the potential for serious adverse reactions in breastfed infants from carboplatin/paclitaxel and nivolumab, women are advised not to breast-feed during treatment with carboplatin/paclitaxel or nivolumab
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* Any prior therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if > 3 years prior to study;
* Any history of active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Uncontrolled diarrhea;
  * Uncontrolled adrenal insufficiency;
  * Transmural myocardial infarction within the last 3 months;
  * Acute bacterial or fungal infection requiring systemic antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
  * Acquired Immune Deficiency Syndrome (AIDS) with CD4+ count < 350 cells per microL; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Women who are breastfeeding and are not willing to discontinue breastfeeding during the trial
* Poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite 2 attempts to improve glucose control by fasting duration and adjustment of medications. Patients with diabetes will preferably be scheduled in the morning and instructions for fasting and use of medications will be provided in consultation with the patients' primary physicians
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Short bursts of steroids of 5-7 days (for COPD exacerbation or other similar indication) are allowed.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to nivolumab or any of its excipients or known hypersensitivity to carboplatin/paclitaxel.
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Received a live vaccine within 30 days of planned start of study therapy.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects screen failed before enrollment
Period: Overall Study
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Started | 26
Completed | 13
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated using the Kaplan-Meier method. Evaluated using imaging and clinical exams
Time Frame: Up to 2 years after completion of study treatment
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
percentage of patients | 65 [46 to 79]

2. Secondary Outcome: Proportion of Patients Who Progressed in Any Location
Description: To characterize patterns of failure, investigators will summarize the proportion of patients who progressed in any location and whether the first progression was local, regional, distant or in multiple locations.
Time Frame: Up to 2 years after completion of study treatment
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
percentage of patients | 15 [7 to 33]

3. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the Kaplan-Meier method
Time Frame: 2 years after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
Participants | 26

4. Secondary Outcome: Incidence of Acute Toxicity
Description: Toxicity evaluation per CTCAE v 5.0
Time Frame: at 1 month post chemoradiation
Measure: Number; unit: Number of Incidents Occurred
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
Number of Incidents Occurred
  Pain- Grade 1 | 39
  Pain- Grade 2 | 40
  Pain- Grade 3 | 1
  Dysphagia- Grade 1 | 26
  Dysphagia- Grade 2 | 29
  Dysphagia- Grade 3 | 11
  Oral Mucositis- Grade 1 | 21
  Oral Mucositis- Grade 2 | 50
  Oral Mucositis- Grade 3 | 6
  Dermatitis- Grade 1 | 33
  Dermatitis- Grade 2 | 31
  Dermatitis- Grade 3 | 9
  Xerostomia- Grade 1 | 65
  Xerostomia- Grade 2 | 9
  Xerostomia- Grade 3 | 0

5. Secondary Outcome: Incidence of Late Toxicity
Description: Toxicity evaluation per CTCAE v 5.0
Time Frame: 12 months post chemoradiation
Measure: Number; unit: Number of Incidents Occurred
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
Number of Incidents Occurred
  Pain- Grade 1 | 15
  Pain- Grade 2 | 0
  Pain- Grade 3 | 0
  Dysphagia- Grade 1 | 22
  Dysphagia- Grade 2 | 4
  Dysphagia- Grade 3 | 1
  Oral Mucositis- Grade 1 | 0
  Oral Mucositis- Grade 2 | 0
  Oral Mucositis- Grade 3 | 0
  Dermatitis- Grade 1 | 0
  Dermatitis- Grade 2 | 0
  Dermatitis- Grade 3 | 0
  Xerostomia- Grade 1 | 60
  Xerostomia- Grade 2 | 1
  Xerostomia- Grade 3 | 0

6. Secondary Outcome: Correlation of Mid-treatment FDG-PET Scans With Post-treatment PET-CT.
Description: Correlation of metabolic image uptake data on mid-treatment FDG-PET scans performed between fractions 8-12 with standard 12 week post-treatment PET-CT. The number of patients with midtreatment ≥50% decrease of MTV2.5 from baseline.
Time Frame: 12 weeks after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
Number analyzed (Participants) | 26
Participants | 13

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 100 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 3.5 year period.
Arm/Group | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy (N=26)
Allergic reaction (Immune system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Encephalitis infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 2 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Failure to thrive in adult
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, Carboplatin/Paclitaxel, Radiotherapy (N=26)
Alanine aminotransferase increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 17 (18)
Dehydration (Metabolism and nutrition disorders) | 14 (15)
Dermatitis radiation (Injury, poisoning and procedural complications) | 23 (35)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 24 (30)
Dysgeusia (Nervous system disorders) | 25 (36)
Dysphagia (Gastrointestinal disorders) | 9 (13)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Esophageal pain (Gastrointestinal disorders) | 9 (15)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 18 (22)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphedema (Vascular disorders) | 4 (4)
Lymphocyte count decreased (Investigations) | 6 (8)
Mucositis oral (Gastrointestinal disorders) | 25 (48)
Nausea (Gastrointestinal disorders) | 21 (28)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 9 (16)
Pain (General disorders) | 5 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Shingles (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrush (Infections and infestations) | 9 (10)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weight loss (Investigations) | 20 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03829722/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03829722/ICF_001.pdf